CLINICAL TRIAL: NCT02609737
Title: Theranostics of Radiolabeled Somatostatin Antagonists 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11 in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-161
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-12

CONDITIONS: Neuroendocrine Tumors
Keywords: Radiolabeled Somatostatin Antagonists; 68Ga-DOTA-JR11; 177Lu-DOTA-JR11; Pet scan; CT scan; 15-161
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 177Lu-DOTA-JR11

ARMS (1):
- 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11 (Experimental): Pts get a PET/CT study with approx.150-200 MBq of 68Ga-DOTA-JR11. Lesions with focal radiotracer uptake not explained by physiologic sstr2 expression will be interpreted as metastatic disease. If 68Ga-DOTA-JR11 uptake by metastases with a diameter of more than 2 cm is less than the physiologic radiotracer uptake by the liver, no further imaging & therapy will be performed as part of the study, as it is unlikely that pts with this low radiotracer uptake will benefit from PRRT (2). All other pts will undergo a dosimetric study with 1850 MBq (less than 100 μg peptide) of 177Lu-DOTA-JR11. Results of the dosimetry study, will determine the balance of activity of 177Lu-DOTA-JR11 that can be administered without exceeding the radiation dose limits. This activity will be split into 2 equal amounts to be delivered in 2 cycles, approximately 3 months apart. After each therapy cycle, pts will be followed clinically for 3 months.
  Interventions: Device: PET/CT Imaging; Radiation: 68Ga-DOTA-JR11; Radiation: 177Lu-DOTA-JR11

INTERVENTIONS:
Device: PET/CT Imaging
Radiation: 68Ga-DOTA-JR11
Radiation: 177Lu-DOTA-JR11

SUMMARY:
This study has 3 steps and not everyone will have all 3 steps done. The overall goals are to see if a new experimental drug is safe to image (step 1) and treat neuroendocrine tumors (step 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Adults ≥ 18 years old
* Histologically or cytologically confirmed metastatic and/or unresectable progressive, well differentiated carcinoid or pancreatic NET carcinoids
* Progressive metastatic disease defined by one of the following, occurring within 6 months of study entry:

  * At least a 20% increase in radiologically or clinically measurable disease
  * Appearance of any new lesion
  * Symptomatic disease (including worsening hormonal symptoms or symptoms related to tumor burden)
* Measurable disease as defined by RECIST 1.1.
* At least one metastasis must show uptake of 111In-DTPA-octreotide on SPECT that is higher than the physiologic radiotracer uptake by the liver
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3.0 x 109/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelets ≥ 200 x 10^9/L
  * Total bilirubin ≤ 1.25 x Upper Limit Normal (ULN)
  * AST (SGOT)/ ALT(SGPT) ≤ 2.5 x ULN with liver metastases
  * Alkaline phosphatase < 2 x ULN (if known liver or bone disease)
  * Serum albumin > 30 g/L, or serum albumin = 30 g/L but normal prothrombin time
  * Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) calculated CrCl ≥ 60 mL/min/1.73m^2
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Previous local therapy (e.g., chemoembolization or bland embolization) is allowed if completed > 6 weeks prior to study entry. For such patients, there must be either progression of measurable disease documented within the treatment field, or measurable progressive disease outside the treatment field prior to study entry.
* Previous chemotherapy and/or investigational agents are allowed if completed > 4 weeks prior to study entry (> 6 weeks if last regimen contained bis-chloroethyl nitrosourea (BCNU) or mitomycin C). For patients who received systemic therapy prior to study entry, there must be documented progression of measurable disease since receiving systemic therapy prior to study entry.
* Patients must not have disease that is currently amenable to surgery. Prior surgery is allowed no less than 6 weeks prior to study entry.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-DOTA-JR11 as assessed from medical records
* Life expectancy < 6 months as assessed by the treating physician.
* Treatment with short-acting somatostatin analogs less than 3 days and Sandostatin® depot injection less than 5 weeks before scanning and treatment
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or breastfeeding
* Toxicities from prior therapies that have not resolved to grade 1 or grade 0
* Known CNS metastases and/or carcinomatous meningitis
* Active malignancy of metastatic potential other than the known carcinoid or pancreatic NET within the past three years
* >20% bone marrow external beam radiotherapy and/or previous radioisotope therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bodei, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 58 [22 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: according to RECIST 1.1 and median progression-free and overall survival will be estimated and reported with 95% confidence intervals
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11
Number analyzed (Participants) | 20
Participants
  Complete Response | 1
  Partial Response | 8
  Stable Disease | 8
  Progression of Disease | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11
All-Cause Mortality (participants affected / at risk) | 11/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11 (N=20)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 68Ga-DOTA-JR11 and 177Lu-DOTA-JR11 (N=20)
Alopecia (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema (face) (General disorders) | 1
Edema (limbs) (General disorders) | 2
Mucositis (oral) (Gastrointestinal disorders) | 1
Asthenia (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT02609737/Prot_SAP_000.pdf